CLINICAL TRIAL: NCT07190196
Title: A Randomized, Phase 3, Double-blind, 52-week Study to Evaluate the Efficacy and Safety of Rilzabrutinib (SAR444671) Compared to Placebo in Adult Participants With Active IgG4-related Disease
Brief Title: A 52-week Study of Rilzabrutinib Efficacy and Safety Compared to Placebo in Adults Diagnosed With IgG4-related Disease
Acronym: RILIEF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17359; U1111-1316-0266 (Registry Identifier: WHO ICTRP); 2025-521398-15 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Immunoglobulin G4 Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rilzabrutinib (Experimental): Rilzabrutinib
  Interventions: Drug: Rilzabrutinib; Drug: Glucocorticoid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Drug: Glucocorticoid

INTERVENTIONS:
Drug: Rilzabrutinib — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: SAR444671
  Arms: Rilzabrutinib
Drug: Placebo — Pharmaceutical form:Tablet-Route of administration:Oral
  Arms: Placebo
Drug: Glucocorticoid — Pharmaceutical form:Tablet, solution, suspension formulations according to local standard practices-Route of administration:Oral

SUMMARY:
This is a Phase 3, parallel group, 2-arm, randomized, double blind, placebo-controlled, 52-week treatment study to assess the efficacy and safety of rilzabrutinib as a treatment for adult patients with active IgG4-RD.

The purpose of this study is to measure time to IgG4-RD clinical disease flare, and other relevant efficacy endpoints including flare-free rate, control of IgG4-RD disease activity, use of GC rescue and safety parameters such as treatment-emergent adverse events, clinical laboratory values and electrocardiograms (ECG) in participants aged 18 years and above, diagnosed with IgG4-RD and treated with rilzabrutinib tablets over a 52-week placebo-controlled period.

Study details include:

The study duration will be up to 60 weeks, including a 4 to 6-week screening period, a 52-week double blind treatment period, and 2 weeks of follow up (plus an optional OLE of 108 weeks).

The number of visits will be 16 (plus an optional 9 visits during the OLE).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an adjudicated clinical diagnosis of IgG4-RD
* Participants meeting Step 1 Entry criteria of 2019 ACR/EULAR classification criteria for IgG4-RD and Total inclusion points are ≥20
* Participants with active disease at screening in at least one organ system, excluding lymph nodes, as an IgG4-RD Responder Index total activity score ≥ 2
* Participants with history or current involvement of at least 1 organ/site (excluding lymph nodes) affected with IgG4-RD.
* Participants with active IgG4-RD controlled for at least 2 weeks while on a stable dose of GC.
* Participants willing to taper off GC after starting IMP.
* Participants willing and able to participate in repeated study protocol mandated or clinically indicated imaging procedures to assess IgG4-RD such as computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), or ultrasound.
* Participants who have an up-to-date vaccination status as per local guidelines. The last dose of live vaccines should be received at least 30 days before Day 1.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Meet any Step 2 Exclusion criteria from the 2019 ACR/EULAR classification criteria for IgG4-RD.
* History of retroperitoneal fibrosis, sclerosing mesenteritis, fibrosing mediastinitis, or other overwhelmingly fibrotic expression of IgG4-RD that is the sole disease manifestation.
* Active malignancy or history of malignancy within 5 years before Day 1, except completely treated in situ carcinoma of the cervix, completely treated, and resolved nonmetastatic squamous or basal cell carcinoma of the skin.
* Known or suspected immunodeficiency, including history of invasive opportunistic infections (eg, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency or prolonged duration suggesting an immune compromised status, as judged by the Investigator.
* History of serious infections with the potential for recurrence (as judged by the Investigator), with less than 4 weeks interval between resolution of serious infection and first dose of study drug, or currently active moderate to severe infection at Screening (Grade 2 or higher).
* Current or chronic history of liver disease unrelated to IgG4-RD.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, bariatric surgery, or significant bowel resection that would preclude adequate rilzabrutinib/placebo absorption.
* History of solid organ transplant.
* Planned major surgical procedure during the participation in this study.
* History of drug abuse within the previous 12 months.
* Alcoholism or excessive alcohol use, defined as regular consumption of more than approximately 3 standard drinks per day.
* Prior participation in any rilzabrutinib studies or other BTK inhibitor studies.
* History of treatment with an investigational drug within 6 months or 5 half-lives of the investigational drug, whichever is longer.
* Laboratory abnormalities at the screening visit identified by the central laboratory The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-06-28 (Estimated); Study Completion 2030-12-25 (Estimated)

PRIMARY OUTCOMES:
Time to first adjudicated clinical disease flare treated by the investigator during the Blinded Treatment period | Until Week 52
  The Adjudication Committee will include internationally recognized independent experts in diagnosis and management of patients with IgG4-RD, blinded to participant, investigator, and site identifiers

SECONDARY OUTCOMES:
Percentage of participants without IgG4-RD adjudicated clinical disease flare and off glucocorticoids and immunomodulators | At Week 52
Percentage of participants without IgG4-RD adjudicated clinical disease flare and off glucocorticoids | At Week 52
Annualized rate of clinical disease flares | At Week 52
Change in IgG4-RD RI total activity scores from baseline to Week 52 | From baseline to Week 52
Percent change in IgG4-RD RI total activity scores form baseline to Week 52 | From baseline to Week 52
Change in IgG4-RD RI total activity scores from baseline to Week 12 | From baseline to Week 12
Proportion of participants with reduction of ≥2 points from the baseline IgG4-RD RI total activity score | At Week 12, Week 24, and Week 52
Proportion of participants in complete remission | At Week 52
  Defined by an IgG4-RD RI total activity score = 0 or absence of evident disease activity assessed by the Investigator
Cumulative glucocorticoid dose for treatment of IgG4-RD | At Week 52
Proportion of participants with potentially clinically significant abnormalities in laboratory tests, vital signs, and electrocardiograms in the Safety Population | Until Week 160
Proportion of participants with TEAEs, AESIs, SAEs in the Safety Population | Until Week 160

CONTACTS AND LOCATIONS:
Locations (40):
- United States (7):
  - San Jose Clinical Trials- Site Number : 8400016, San Jose, California
  - Life Clinical Trials- Site Number : 8400002, Margate, Florida
  - Primeway Clinical Research Group- Site Number : 8400019, Fayetteville, Georgia
  - Paramount Medical Research & Consulting, LLC- Site Number : 8400018, Middleburg Heights, Ohio
  - Stryde Research- Site Number : 8400011, Plano, Texas
  - Epic Medical Research (Red Oak)- Site Number : 8400003, Red Oak, Texas
  - Velocity Clinical Research Seattle- Site Number : 8400005, Seattle, Washington
- Investigational Site Number : 0320004, Buenos Aires, Argentina
- Investigational Site Number : 1240001, Sherbrooke, Quebec, Canada
- Chile (5):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Concepción, Región del Biobío
  - Investigational Site Number : 1520002, Santiago
- China (6):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560012, Chengdu
  - Investigational Site Number : 1560010, Hangzhou
  - Investigational Site Number : 1560003, Shijiazhuang
  - Investigational Site Number : 1560011, Wuhan
  - Investigational Site Number : 1560009, Yantai
- Israel (3):
  - Investigational Site Number : 3760003, Nahariya
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760005, Tel Aviv
- Italy (2):
  - AOU Meyer IRCCS-Site Number : 3800003, Florence, Tuscany
  - Centro Ricerche Cliniche di Verona s.r.l. c/o Policlinico G.B.Rossi-Site Number : 3800002, Verona, Veneto
- Japan (4):
  - Investigational Site Number : 3920010, Kobe, Hyōgo
  - Investigational Site Number : 3920002, Kahoku-gun, Ishikawa-ken
  - Investigational Site Number : 3920005, Nagaoka-shi, Niigata
  - Investigational Site Number : 3920004, Kitakyushu
- Netherlands (2):
  - Investigational Site Number : 5280002, Groningen
  - Investigational Site Number : 5280001, Rotterdam
- Poland (2):
  - Investigational Site Number : 6160001, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160003, Gdansk, Pomeranian Voivodeship
- South Korea (2):
  - Investigational Site Number : 4100002, Suwon, Gyeonggi-do
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (3):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Madrid
- Sweden (2):
  - Investigational Site Number : 7520001, Stockholm
  - Investigational Site Number : 7520002, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17359 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26866&tenant=MT_SNY_9011